CLINICAL TRIAL: NCT01573611
Title: Examining the Impact of Grape Consumption on Brain Metabolism and Cognitive Function in Patients With Mild Cognitive Impairment
Brief Title: Impact of Grape Consumption on Brain Metabolism and Cognitive Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Daniel H. Silverman, Professor, Molecular and Medical Pharmacology, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 11002966
Record Dates: First submitted 2012-04-05; First posted 2012-04-09 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Mild Cognitive Impairment
Keywords: mild cognitive impairment; dementia; positron emission tomography (PET); F-18 Fluorodeoxyglucose (FDG); cerebral metabolism; dietary supplement
MeSH Terms: conditions — Cognitive Dysfunction; Dementia | interventions — whole grape extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Grape Powder (Experimental)
  Interventions: Dietary Supplement: Grape Powder
- Placebo Powder (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo Powder

INTERVENTIONS:
Dietary Supplement: Grape Powder — 36 g of grape powder to be taken twice/day (total of 72 g/day) for 6 months
  Arms: Grape Powder
Dietary Supplement: Placebo Powder — 36 g of placebo powder to be taken twice/day (total of 72 g/day) for 6 months
  Arms: Placebo Powder

SUMMARY:
Constituents of grapes have been studied for their antioxidant, anti-inflammatory, and anticarcinogenic properties. In the past decade, there has been emerging evidence regarding a potential role for grapes in slowing cognitive decline and other effects of aging. Furthermore, evidence has been obtained in vivo that supplementation of aged rats with grape seed extract improves cognitive performance. Despite the promising accumulating data supporting the use of grapes as a safe and effective strategy for delaying the incidence of dementia, it remains unclear how grape intake would be useful with respect to factors such as dose schedule or stage of dementing illness. In general, well-controlled experimental data obtained in human subjects is in need of much further development. The investigators aim to measure effects of grape intake on cerebral metabolism and cognitive function, and to determine whether initial patterns, and magnitude of change, of cerebral metabolism assessed by positron emission tomography (PET) can serve respectively as a predictor of, and biomarker for, the magnitude of cognitive changes resulting from intake of grapes.

DETAILED DESCRIPTION:
People experiencing mild cognitive changes represent an epidemiologically major segment of the geriatric patient population. Numerous studies have been carried out to study the benefits of grapes associated with dementia and Alzheimer's disease (AD). In the present proposal, the investigators aim to determine 1) whether cognitive and regional cerebral metabolic changes associated with grape powder use can be identified, 2) if the presence and magnitude of therapeutic responses to grape in patients having mild cognitive decline can be predicted by particular patterns of regional brain metabolism, and 3) for any changes identified, the magnitude of those changes that correlate with the magnitude of the changes noted in the neuropsychologic parameters will be examined, which might be useful as an objective biomarker for therapeutic effect. A total of 12 patients suffering from documented decline of cognitive function (in the absence of overt dementia) will be studied. In this placebo-controlled, double-blinded study, the 12 recruited subjects who have met the screening criteria will be randomized to receive 72 g of grape powder per day or placebo. The subjects will undergo a baseline brain PET study with the radiotracer [F - 18] fluorodeoxyglucose (FDG). In addition, neuropsychological assessments will be performed at baseline and six months after initiation of therapy. Follow-up PET scans will also be obtained at six months to assess the changes in metabolism occurring with each therapy regimen.

ELIGIBILITY:
Inclusion Criteria:

* Cognitive deficit and/or personality change is present, as observable by physician and/or close contact(s) of the patient; or in the absence of this, the patient provides a clear history of decline which the patient's physician deems to be reliable.
* If history or neurologic exam reveals findings suspicious for stroke, tumor, bleed, ictal activity, or hydrocephalus, then CT/MRI and appropriate neurological or neurosurgical consultation must have been obtained.
* Standard history, physical, and laboratory screen have been performed to identify possible presence of depression, substance abuse, malnourishment, medication effects and interactions, cardiopulmonary compromise, electrolyte/calcium imbalance, anemia, hypoxemia, infection, thyroid dysfunction, renal dysfunction, hepatic dysfunction, or glucose dysregulation.
* Any positive findings revealed in 2) or 3) above have been appropriately treated, wherever possible, but cognitive/behavioral deficit persists post-therapy.

Exclusion Criteria:

* Subjects under age 65 will not be recruited, in order to enhance the clinical relevance of the project by focusing on the age groups in whom serious concerns about early signs and symptoms of senile onset dementia are most typically emerging.
* Already diagnosed with Alzheimer's disease or other cause of dementia
* Cognitive dysfunction has impaired subject's ability to perform activities of daily living.
* Present or past history of thyroid disease (due to effects of both the disease and thyroid hormone replacement therapy on brain metabolism that we and others have begun to identify, but which remain incompletely characterized.)
* Claustrophobia or metal in body or other condition that would preclude PET or MRI from being acquired, or visual, auditory or motor deficits that would preclude accurate neuropsychological testing.
* Currently receiving medication used specifically to treat Alzheimer's disease or other dementia-related disorder

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-04; Primary Completion 2013-04 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in neuropsychological (cognitive, functional) test results | baseline and 6 months
Change from baseline in regional cerebral metabolism | baseline and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Daniel H. Silverman, MD, Ph.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Medical Center, Los Angeles, California, United States